CLINICAL TRIAL: NCT01796340
Title: Cue Exposure Training for Overweight Children
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient number of participants
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Maastricht University (Other); Netherlands Organisation for Scientific Research (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: METC 13-2-009; NWO (Other Grant/Funding Number: Vici grant 453.10.006, awarded to Anita Jansen)
Record Dates: First submitted 2013-02-20; First posted 2013-02-21 (Estimated); Last update posted 2015-10-15 (Estimated); Status verified 2014-10

CONDITIONS: Overweight; Obesity
Keywords: cue exposure; childhood; overeating; overweight; obese; treatment
MeSH Terms: conditions — Overweight; Obesity; Hyperphagia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Food cue exposure (Experimental)
  Interventions: Behavioral: Food cue exposure
- Psycho-education (Active Comparator)
  Interventions: Behavioral: Psycho-education

INTERVENTIONS:
Behavioral: Food cue exposure — Participants will be exposed to several kinds of their favorite food. The aim of this exposure is to increase the food cravings as much as possible.
  Arms: Food cue exposure
Behavioral: Psycho-education — General information about nutrients, calories, exercise and the energy balance will be provided. In addition, psychological problems that accompany overweight will be discussed.
  Arms: Psycho-education

SUMMARY:
The primary objective of the study is to investigate the effectiveness of two intensive two-session trainings, the conventional psycho-education and food cue exposure, on eating in the absence of hunger, binge eating and Body Mass Index (BMI) change in overweight/ obese children.

ELIGIBILITY:
Inclusion Criteria:

* Being a patient in the Maastricht University Medical Center COACH unit for obese children and adolescents.
* Overweight, according to the sex and age specific cut-off point for overweight in children, as defined by Cole and colleagues (2000).
* Age: 12 - 18 years

Exclusion Criteria:

* Not being overweight (anymore, due to weight loss)
* Not able to speak and/or write Dutch

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 14 (Actual)
Dates: Start 2014-01; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Eating in the absence of hunger | 2 - 3 months
  Self-reported & behaviourally measured eating in the absence of hunger
Binge eating | 2 - 3 months
  Self-reported binge eating

SECONDARY OUTCOMES:
Cue reactivity | 2 - 3 months
  Reactivity to food related cues, measured by food cravings and salivary responses
Self-control and self-esteem | 2 - 3 months
  Self-reported self-control and self-esteem
Dietary restraint, and eating, weight and shape concerns | 2 - 3 months
  Self-reported dietary restraint, and eating, weight and shape concerns
BMI change | 2 - 3 months
  Body Mass Index change

OTHER OUTCOMES:
Self-reported expectation and evaluation of intervention | 2 - 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Anita Jansen, Professor, Principal Investigator — Maastricht University
Locations (1):
- Maastricht University Medical Centre (MUMC+), Maastricht, Limburg, Netherlands

REFERENCES:
- [Background] Jansen A, Van den Hout MA, De Loof C, Zandbergen J, Griez E. A case of bulimia successfully treated by cue exposure. J Behav Ther Exp Psychiatry. 1989 Dec;20(4):327-32. doi: 10.1016/0005-7916(89)90064-5. PMID 2576871
- [Background] Jansen A, Broekmate J, Heymans M. Cue-exposure vs self-control in the treatment of binge eating: a pilot study. Behav Res Ther. 1992 May;30(3):235-41. doi: 10.1016/0005-7967(92)90069-s. PMID 1586360
- [Background] Jansen A. A learning model of binge eating: cue reactivity and cue exposure. Behav Res Ther. 1998 Mar;36(3):257-72. doi: 10.1016/s0005-7967(98)00055-2. PMID 9642846
- [Background] Toro J, Cervera M, Feliu MH, Garriga N, Jou M, Martinez E, Toro E. Cue exposure in the treatment of resistant bulimia nervosa. Int J Eat Disord. 2003 Sep;34(2):227-34. doi: 10.1002/eat.10186. PMID 12898559
- [Background] Martinez-Mallen E, Castro-Fornieles J, Lazaro L, Moreno E, Morer A, Font E, Julien J, Vila M, Toro J. Cue exposure in the treatment of resistant adolescent bulimia nervosa. Int J Eat Disord. 2007 Nov;40(7):596-601. doi: 10.1002/eat.20423. PMID 17607695
- [Background] Boutelle KN, Zucker NL, Peterson CB, Rydell SA, Cafri G, Harnack L. Two novel treatments to reduce overeating in overweight children: a randomized controlled trial. J Consult Clin Psychol. 2011 Dec;79(6):759-71. doi: 10.1037/a0025713. PMID 22122291